CLINICAL TRIAL: NCT06846918
Title: HIIT Vs Snack Exercises on the Academic Stress of University Students: a Randomized Controlled Trial
Brief Title: HIIT Vs Snack Exercises on the Academic Stress of University Students
Acronym: SHARP-Stress
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Metropolitana de Ciencias de la Educacion (Other)
Responsible Party: Principal Investigator, Mauricio Inostroza Mondaca, Principal Investigator, Universidad Metropolitana de Ciencias de la Educacion
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07-2025-ID DIUMCE; DIUMCE 07-2025-ID (Other Grant/Funding Number: Universidad Metropolitana de Ciencias de la Educación)
Record Dates: First submitted 2025-02-20; First posted 2025-02-26 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Mental Health; Mental Health Care; Physical Inactivity; Sedentary Behaviors; Cardiovascular Health
Keywords: High-intensity Interval Training; Snack Exercises; Academic Stress; Mental Health Well-being
MeSH Terms: conditions — Psychological Well-Being; Sedentary Behavior | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High-intensity Interval Training Group (Active Comparator)
  Interventions: Behavioral: High-Intensity Interval Training
- Snack Exercises Group (Experimental)
  Interventions: Behavioral: Exercise Snacks Protocol
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: High-Intensity Interval Training — The high-intensity interval training (HIIT) protocol will run for 12 weeks, with two weekly sessions, totaling 24 sessions. Each 20-minute session will follow a group-based circuit format with functional exercises (e.g., jogging, jumping jacks, step-ups). High-intensity phases will be performed at maximum effort, while moderate-intensity phases will be maintained at a Borg scale rating of 4-6.
  Training will amount to 40 minutes per week. The intensity ratio will progress over time:
  * Weeks 1-4: 15 sec high / 60 sec moderate (1:4)
  * Weeks 5-8: 15 sec high / 45 sec moderate (1:3)
  * Weeks 9-12: 15 sec high / 30 sec moderate (1:2)
  * Weeks 13-16: 15 sec high / 15 sec moderate (1:1)
  This progressive structure ensures gradual adaptation while maximizing effectiveness.
  Arms: High-intensity Interval Training Group
Behavioral: Exercise Snacks Protocol — The exercise snack protocol will last for 12 weeks, with sessions held twice a week, totaling 24 sessions. The exercise snacks will amount to 40 minutes per week, divided across the five weekdays. Participants will be required to perform 4 minutes of functional exercises (e.g., jogging in place, jumping jacks in place, modified burpees in place, etc.) in both the morning (AM) and evening (PM), completing a total of 8 minutes per day. The exercises must be performed at high intensity, with a score of >8 on a modified Borg scale.
  Arms: Snack Exercises Group

SUMMARY:
Mental health among Chilean university students has steadily deteriorated since 2020. One of the factors associated with mental health is the academic workload that comes with transitioning from high school to higher education, which may lead to an increase in stress levels due to university life referred to as academic stress. Academic stress has been linked to multiple negative outcomes in university students, such as a lower quality of life, as well as cardiovascular risk markers, including body composition (e.g., higher fat percentage), muscle function, aerobic capacity, and physical activity levels. Academic stress affecting more than 50% of university students represents a health issue that needs to be addressed, not only because it can lead to chronic stress, but also because it increases cardiovascular risk in a Chilean population where more than 10,000,000 people are overweight, obese, or have insufficient physical activity levels.

Academic stress and its associated complications represent a prevalent health issue among university students. It is essential to implement interventions that help reduce academic stress while also counteracting its negative effects on quality of life, body composition, muscle function, aerobic capacity, and physical activity levels.

Cost-effective tools, both in terms of financial resources and time, are needed. From this perspective, physical exercise meets both requirements, as it is inexpensive to implement and there are various protocols such as high-intensity interval training and "exercise snacks" that can require less than 40 minutes per week while providing beneficial effects on academic stress, body composition muscle function, aerobic capacity, and physical activity levels in university students.

Expanding the body of evidence on these different training protocols would allow us to address multiple issues simultaneously. The primary one is academic stress and its related consequences, but also to generate new evidence on aspects not yet covered in the current literature, such as the impact on university students' quality of life, and to provide an accessible treatment tool for the future. Importantly, implementing these short-duration programs would also enable students to maintain their academic responsibilities, as the proposed protocols require no more than 40 minutes per week (<10 minutes per day). Finally, these programs could be implemented within university facilities, which, in the long term, could become a permanent tool for improving students' university experience.

DETAILED DESCRIPTION:
he mental health of Chilean university students has deteriorated since the COVID-19 pandemic. Academic factors (e.g., workload pressure or fear of poor performance) play a significant role in the development of mental health disorders in university students. One of the most frequently mentioned conditions among Chilean university students is stress, with 56% of students experiencing some form of stress, ranging from mild to extreme. Importantly, academic stress can be a predictor of chronic stress in university students. Therefore, it is essential to manage students' stress levels, as stress is associated with various negative effects on quality of life, body composition, and physical activity levels.

Specifically, a systematic review study found a negative association between academic stress and quality of life in university students. Similarly, higher academic stress scores are associated with a higher body mass index and fat percentage. Likewise, university students with obesity exhibit higher levels of academic stress. Additionally, higher levels of academic stress are linked to lower levels of physical activity. Consequently, the presence of academic stress has a detrimental effect on quality of life, body composition, and physical activity levels. Interestingly, individuals who do not meet adequate physical activity levels also show poorer muscle function and aerobic capacity. Thus, academic stress is involved in both the mental and physical health of university students.

It has been shown that engaging in vigorous physical activity can reduce academic stress among university students. This presents an interesting opportunity to improve the previously mentioned aspects negatively affected by academic stress. Unfortunately, 75.1% of university students report that lack of time is the main reason for not engaging in physical activity. Therefore, it is crucial to propose time-efficient physical activity protocols. In this regard, high-intensity interval training (HIIT) and exercise snack protocols meet the criteria of high intensity and time efficiency. As a result, they could serve as an effective way to promote higher physical activity levels among university students, thereby reducing the negative effects of academic stress on both mental and physical health.

There is some evidence supporting the benefits of high-intensity interval training for reducing stress in university students. Additionally, HIIT protocols have demonstrated positive effects on body composition, leading to a reduction in body fat percentage and visceral adipose tissue, which is closely linked to the development of cardiovascular diseases. Therefore, this type of training protocol could contribute to improvements in cardiovascular risk among university students. Similarly, these training protocols enhance aerobic capacity and muscle function, variables that are also found to be altered in the university population. Interestingly, to the best of our knowledge, no concrete benefits of HIIT protocols on university students' quality of life have been reported. Therefore, this would be a significant aspect of our research, as quality of life is a variable that tends to decline in this population.

Exercise snacks are a more novel tool for achieving health goals in the population, with their main characteristic being the short duration of training intervals (<10 minutes per day in total). The primary goal of this type of training is to break sedentary behavior and increase daily physical activity levels in the population in which they are implemented. Given the high levels of sedentary behavior and low physical activity levels observed in university students, this type of training could serve as a strategy to reduce sedentary behavior and increase physical activity levels. Interestingly, there is evidence supporting the benefits of exercise snacks in improving aerobic capacity, muscle function, and body composition variables that, as previously mentioned, are or could be negatively affected by academic stress in university students. Therefore, implementing a training program of this nature would be beneficial for university students.

Similarly, the application of exercise snack protocols has been associated with higher enjoyment compared to HIIT protocols, likely due to their shorter duration. Finally, to the best of our knowledge, there is limited evidence regarding the effects of exercise snack protocols on academic stress and quality of life in university students. Thus, generating evidence on these variables in university students is crucial.

Therefore, the objective of this study is to determine the effects of a high-intensity interval training protocol versus an exercise snack protocol on academic stress, quality of life, body composition, muscle function, and aerobic capacity in university students.

ELIGIBILITY:
Inclusion Criteria:

* University students from the 1st to 4th year at the Metropolitan University of Education Sciences and Silva-Henriquez Catholic University

Exclusion Criteria:

* High level of physical activity classification in the GPAQ questionnaire.
* Musculoskeletal conditions that prevent normal physical activity.
* Cardiac disease that contraindicates high-intensity exercise.
* Diagnosed mental health condition.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Academic Stress Levels | T0 (before the training protocol) and T12 (after 12 weeks of training).
  It will be measured using the SISCO II questionnaire, validated in the Chilean population, with items rated on a Likert scale from 1 to 5. The questionnaire consists of five dimensions: stressors, physical and psychological reactions, social behavior reactions, coping strategies, and total reaction.

SECONDARY OUTCOMES:
Quality of Life Levels | T0 (before the training protocol) and T12 (after 12 weeks of training).
  It will be measured using the SF-36 questionnaire, which assesses eight dimensions: physical function, physical role, bodily pain, general health, vitality, social function, emotional role, and mental health. Scores are obtained through a Likert-type scale, which must be transformed to a 0-100 scale, where 0 represents the worst performance and 100 the best. The questionnaire has been validated in Spanish-speaking populations.
Physical Activity Levels | T0 (before the training protocol) and T12 (after 12 weeks of training).
  The Global Physical Activity Questionnaire (GPAQ) assesses physical activity across three domains: work-related activity, transportation activity, and recreational activity. It also includes a section on sedentary behavior. The questionnaire measures the frequency and duration of moderate and vigorous physical activity in each domain, providing a comprehensive overview of an individual's physical activity levels. In the Chilean population, the GPAQ has been validated, with studies confirming its reliability in national health surveys.
Sedentary Behaviour Levels | T0 (before the training protocol) and T12 (after 12 weeks of training)
  The Global Physical Activity Questionnaire (GPAQ) assesses physical activity across three domains: work-related activity, transportation activity, and recreational activity. It also includes a section on sedentary behavior. The questionnaire measures the frequency and duration of moderate and vigorous physical activity in each domain, providing a comprehensive overview of an individual's physical activity levels. In the Chilean population, the GPAQ has been validated, with studies confirming its reliability in national health surveys. Additionally, research has shown that the single-question measure of sedentary behavior within the GPAQ is a valid tool for assessing sedentary time in Chilean adults.
Upper Body Muscle Strength | T0 (before the training protocol) and T12 (after 12 weeks of training)
  A 10RM test will be conducted to assess upper limb strength (bench press). The Epley formula will be used to estimate 1RM from the 10RM test.
Lower Body Muscle Strength | T0 (before the training protocol) and T12 (after 12 weeks of training)
  A 10RM test will be conducted to assess lower limb strength (squat). The Epley formula will be used to estimate 1RM from the 10RM test
Aerobic Capacity | T0 (before the training protocol) and T12 (after 12 weeks of training).
  A maximal oxygen consumption test will be conducted to estimate the participants' aerobic capacity.
Body Weight | T0 (before the training protocol) and T12 (after 12 weeks of training).
  Will be measured using a scale and stadiometer SECA ®.
Height | T0 (before the training protocol) and T12 (after 12 weeks of training).
  Will be measured using a scale and stadiometer SECA ®.
Body Mass Index | T0 (before the training protocol) and T12 (after 12 weeks of training).
  Body mass index (BMI) will be calculated based on the weight and height values.
Waist Circumference | T0 (before the training protocol) and T12 (after 12 weeks of training).
  Waist circumference will be measured using a non-extensible SECA® tape
Waist to Height Ratio | T0 (before the training protocol) and T12 (after 12 weeks of training).
  Will be calculated using the values of height and waist circumference
Skeletal Muscle Mass | T0 (before the training protocol) and T12 (after 12 weeks of training).
  It will be assessed using a bioelectrical impedance analysis (BIA).
Fat mass | T0 (before the training protocol) and T12 (after 12 weeks of training).
  It will be assessed using a bioelectrical impedance analysis (BIA).
Fat Mass Percentage | T0 (before the training protocol) and T12 (after 12 weeks of training).
  It will be assessed using a bioelectrical impedance analysis (BIA).
Visceral Adiposse Tissue Area | T0 (before the training protocol) and T12 (after 12 weeks of training).
  It will be assessed using a bioelectrical impedance analysis (BIA).
Physical Activity Enjoyment | T0 (before the training protocol) and T12 (after 12 weeks of training).
  The Physical Activity Enjoyment Scale will be used to assess the enjoyment of the two different training programs. The questionnaire consists of 16 Likert-type questions and was validated in the Spanish language and presents a Cronbach's Alpha coefficient of 0.85, informing an internal consistency of the scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Metropolitana de Ciencias de la Educación, Metropolitana, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Yes